CLINICAL TRIAL: NCT00940251
Title: Evaluation of Safety and Efficacy of Mersina, an Ayurvedic Formulation: A Double Blind, Placebo Controlled Study in Type 2 Diabetic Patients With Secondary Failure to Oral Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jyoti Clinical and Pathological Laboratory (Other)
Responsible Party: Jayavant M Jain, Jyoti Clinical and Pathological Laboratory
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MER1
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Antihyperglycemic Effect in Type 2 Diabetic Patients With Secondary Failure to Oral Hypoglycemic Agents
Keywords: Ayurvedic formulation; type 2 diabetes mellitus; secondary failure to oral hypoglycemic agents; antidiabetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CORN STARCH (Placebo Comparator)
  Interventions: Drug: Mersina
- Mersina, Diet and exercise (Active Comparator)
  Interventions: Drug: Mersina

INTERVENTIONS:
Drug: Mersina — capsule, 3g/day, 3 months

SUMMARY:
To determine the safety and efficacy of an Ayurvedic formulation, Mersina in type 2 diabetic patients with secondary failure to oral hypoglycemic agents, a randomized double blind, single centre, study of 3 months duration was carried out.

ELIGIBILITY:
Inclusion Criteria:

Secondary failure to Oral Hypoglycemic Agents was diagnosed if the patient had HbA1c levels > 8.5% even after supplementation of maximal dose of a combination of a sulphonylurea (15 mg glybenclamide or 160 mg gliclazide or 15 mg glipizide) and metformin 1500 mg/day.

Exclusion Criteria:

Patients with ketosis, diabetes related complications, hepatic or renal disease, pancreatitis, cardiac problems, uncontrolled hypertension, malnutrition and severe immune deficiency

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
antidiabetic activity | 3 months

SECONDARY OUTCOMES:
Improvement in metabolic, insulin level, HbA1c,kidney and lipid profile | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jyoti Clinical and Pathological Laboratory, Shirpur, Maharashtra, India